CLINICAL TRIAL: NCT06015204
Title: Objective Assessment of Extent of Anesthesia in the 8th Cervical Dermatome Using Photoplethysmographic Amplitude in Patients Undergoing Interscalene Brachial Plexus Block
Brief Title: Assessment of the C8 Dermatomal Block with Photoplethysmographic Amplitude After Interscalene Brachial Plexus Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: JongHae Kim (Other)
Collaborators: Research Institute of Medical Science, Daegu Catholic University (Unknown)
Responsible Party: Sponsor-Investigator, JongHae Kim, Professor, Daegu Catholic University Medical Center
Organization: Daegu Catholic University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 2023-02
Record Dates: First submitted 2023-08-18; First posted 2023-08-29 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2023-09

CONDITIONS: Brachial Plexus Block; Oximetry

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- C5-C6 group (Active Comparator): The C5-to-C6 nerve roots and supraclavicular nerves are blocked with 25 ml of 0.75% ropivacaine under ultrasound guidance.
  Interventions: Procedure: Interscalene brachial plexus block targeting the C5-to-C6 nerve roots
- C5-C8 group (Experimental): The C5-to-C8 nerve roots and supraclavicular nerves are blocked with 25 ml of 0.75% ropivacaine under ultrasound guidance.
  Interventions: Procedure: Interscalene brachial plexus block targeting the C5-to-C8 nerve roots

INTERVENTIONS:
Procedure: Interscalene brachial plexus block targeting the C5-to-C6 nerve roots — With the head rotated contralateral to interscalene brachial plexus block (ISBPB), the compactly arranged brachial plexus is visualized lateral to the pulsating subclavian artery under ultrasound guidance. The linear ultrasound transducer is moved cephalad until the C5-to-C8 nerve roots are visualized between the anterior and middle scalene muscles. A block needle is introduced from lateral to medial direction. A nerve root is blocked by placing at least 5 ml of 0.75% ropivacaine around it. The most caudal cervical nerve root (C6 nerve root) is blocked first, and the most cephalad one (C5 nerve root) is blocked last. Then, 3 ml of 0.75% ropivacaine is placed between the scalene and sternocleidomastoid muscles to block the supraclavicular nerves. An equivalent volume of a standard study drug is planned to be used (A total of 25 ml of 0.75% ropivacaine).
  Arms: C5-C6 group
Procedure: Interscalene brachial plexus block targeting the C5-to-C8 nerve roots — With the head rotated contralateral to interscalene brachial plexus block (ISBPB), the compactly arranged brachial plexus is visualized lateral to the pulsating subclavian artery under ultrasound guidance. The linear ultrasound transducer is moved cephalad until the C5-to-C8 nerve roots are visualized between the anterior and middle scalene muscles. A block needle is introduced from lateral to medial direction. A nerve root is blocked by placing at least 5 ml of 0.75% ropivacaine around it. The most caudal cervical nerve root (C8 nerve root) is blocked first, and the most cephalad one (C5 nerve root) is blocked last. Then, 3 ml of 0.75% ropivacaine is placed between the scalene and sternocleidomastoid muscles to block the supraclavicular nerves. An equivalent volume of a standard study drug is planned to be used (A total of 25 ml of 0.75% ropivacaine).
  Arms: C5-C8 group

SUMMARY:
The goal of this clinical trial is to investigate the effectiveness of photoplethysmographic amplitude in assessing the extent of anesthesia in the 8th cervical dermatome in patients undergoing interscalene brachial plexus block (ISBPB). The main question it aims to answer is

* Is there any difference in the post-block changes in photoplethysmographic amplitude measured from the ipsilateral 5th finger (supplied by the 8th cervical nerve root) between ISBPBs targeting the C5-to-C6 nerve roots and the C5-to-C8 nerve roots?
* Do the changes in photoplethysmographic amplitude represent the extent of anesthesia in the 8th cervical dermatome? Participants will receive either ISBPB targeting the C5-to-C6 nerve roots or the C5-to-C8 nerve roots, and then the changes in photoplethysmographic amplitude will be measured from the 5th finger ipsilateral to ISBPB.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status 1 or 2
* Schedule to receive interscalene brachial plexus block for arthroscopic shoulder surgery

Exclusion Criteria:

* Coagulopathy
* Peripheral vascular diseases
* Arrhythmias
* Cardiac conduction abnormalities
* A history of medication affecting cardiac conduction
* Ischemic heart disease
* Hypertension
* Diabetes mellitus
* Thyroid dysfunction
* Other medical conditions affecting autonomic nervous activity
* Infection at the skin area for interscalene brachial plexus block
* Peripheral neuropathy or neurologic sequelae in the upper limb ipsilateral to the surgery
* Allergy to local anesthetics or a history of allergic shock
* Contralateral vocal cord palsy, hemidiaphragmatic paresis/paralysis or pneumo/hemo thorax
* Severe restrictive pulmonary disorder
* Electrolyte imbalance
* Difficulty in communicating with medical personnel
* Patients refusal

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2023-09-13 (Actual); Primary Completion 2024-08-28 (Actual); Study Completion 2024-08-28 (Actual)

PRIMARY OUTCOMES:
Time to achieve 50% of maximum photoplethysmographic amplitude measured from the 5th finger | 25 minutes after the introduction of a block needle
  During the whole study period, the photoplethysmographic waveform obtained from the 1st and 5th fingers ipsilateral to interscalene brachial plexus block is recorded at 100 Hz. The photoplethysmographic amplitude is calculated by subtracting the valley amplitude from the peak amplitude of one heartbeat in photoplethysmographic waveform. Using all the photoplethysmographic amplitudes between 0 and 25 minutes after the introduction of a block needle, a sigmoid Emax model is built. From the model, the time point, when 50% of maximum photoplethysmographic amplitude is achieved, can be derived.

SECONDARY OUTCOMES:
Time to achieve 5% of maximum photoplethysmographic amplitude measured from the 5th finger | 25 minutes after the introduction of a block needle
  During the whole study period, the photoplethysmographic waveform obtained from the 1st and 5th fingers ipsilateral to interscalene brachial plexus block is recorded at 100 Hz. The photoplethysmographic amplitude is calculated by subtracting the valley amplitude from the peak amplitude of one heartbeat in photoplethysmographic waveform. Using all the photoplethysmographic amplitudes between 0 and 25 minutes after the introduction of a block needle, a sigmoid Emax model is built. From the model, the time point, when 5% of maximum photoplethysmographic amplitude is achieved, can be derived.
Time to achieve 10% of maximum photoplethysmographic amplitude measured from the 5th finger | 25 minutes after the introduction of a block needle
  During the whole study period, the photoplethysmographic waveform obtained from the 1st and 5th fingers ipsilateral to interscalene brachial plexus block is recorded at 100 Hz. The photoplethysmographic amplitude is calculated by subtracting the valley amplitude from the peak amplitude of one heartbeat in photoplethysmographic waveform. Using all the photoplethysmographic amplitudes between 0 and 25 minutes after the introduction of a block needle, a sigmoid Emax model is built. From the model, the time point, when 10% of maximum photoplethysmographic amplitude is achieved, can be derived.
Time to achieve 90% of maximum photoplethysmographic amplitude measured from the 5th finger | 25 minutes after the introduction of a block needle
  During the whole study period, the photoplethysmographic waveform obtained from the 1st and 5th fingers ipsilateral to interscalene brachial plexus block is recorded at 100 Hz. The photoplethysmographic amplitude is calculated by subtracting the valley amplitude from the peak amplitude of one heartbeat in photoplethysmographic waveform. Using all the photoplethysmographic amplitudes between 0 and 25 minutes after the introduction of a block needle, a sigmoid Emax model is built. From the model, the time point, when 90% of maximum photoplethysmographic amplitude is achieved, can be derived.
Time to achieve 95% of maximum photoplethysmographic amplitude measured from the 5th finger | 25 minutes after the introduction of a block needle
  During the whole study period, the photoplethysmographic waveform obtained from the 1st and 5th fingers ipsilateral to interscalene brachial plexus block is recorded at 100 Hz. The photoplethysmographic amplitude is calculated by subtracting the valley amplitude from the peak amplitude of one heartbeat in photoplethysmographic waveform. Using all the photoplethysmographic amplitudes between 0 and 25 minutes after the introduction of a block needle, a sigmoid Emax model is built. From the model, the time point, when 95% of maximum photoplethysmographic amplitude is achieved, can be derived.
Time to achieve 99% of maximum photoplethysmographic amplitude measured from the 5th finger | 25 minutes after the introduction of a block needle
  During the whole study period, the photoplethysmographic waveform obtained from the 1st and 5th fingers ipsilateral to interscalene brachial plexus block is recorded at 100 Hz. The photoplethysmographic amplitude is calculated by subtracting the valley amplitude from the peak amplitude of one heartbeat in photoplethysmographic waveform. Using all the photoplethysmographic amplitudes between 0 and 25 minutes after the introduction of a block needle, a sigmoid Emax model is built. From the model, the time point, when 99% of maximum photoplethysmographic amplitude is achieved, can be derived.
Time to achieve 5% of maximum photoplethysmographic amplitude measured from the 1st finger | 25 minutes after the introduction of a block needle
  During the whole study period, the photoplethysmographic waveform obtained from the 1st and 5th fingers ipsilateral to interscalene brachial plexus block is recorded at 100 Hz. The photoplethysmographic amplitude is calculated by subtracting the valley amplitude from the peak amplitude of one heartbeat in photoplethysmographic waveform. Using all the photoplethysmographic amplitudes between 0 and 25 minutes after the introduction of a block needle, a sigmoid Emax model is built. From the model, the time point, when 5% of maximum photoplethysmographic amplitude is achieved, can be derived.
Time to achieve 10% of maximum photoplethysmographic amplitude measured from the 1st finger | 25 minutes after the introduction of a block needle
  During the whole study period, the photoplethysmographic waveform obtained from the 1st and 5th fingers ipsilateral to interscalene brachial plexus block is recorded at 100 Hz. The photoplethysmographic amplitude is calculated by subtracting the valley amplitude from the peak amplitude of one heartbeat in photoplethysmographic waveform. Using all the photoplethysmographic amplitudes between 0 and 25 minutes after the introduction of a block needle, a sigmoid Emax model is built. From the model, the time point, when 10% of maximum photoplethysmographic amplitude is achieved, can be derived.
Time to achieve 50% of maximum photoplethysmographic amplitude measured from the 1st finger | 25 minutes after the introduction of a block needle
  During the whole study period, the photoplethysmographic waveform obtained from the 1st and 5th fingers ipsilateral to interscalene brachial plexus block is recorded at 100 Hz. The photoplethysmographic amplitude is calculated by subtracting the valley amplitude from the peak amplitude of one heartbeat in photoplethysmographic waveform. Using all the photoplethysmographic amplitudes between 0 and 25 minutes after the introduction of a block needle, a sigmoid Emax model is built. From the model, the time point, when 50% of maximum photoplethysmographic amplitude is achieved, can be derived.
Time to achieve 90% of maximum photoplethysmographic amplitude measured from the 1st finger | 25 minutes after the introduction of a block needle
  During the whole study period, the photoplethysmographic waveform obtained from the 1st and 5th fingers ipsilateral to interscalene brachial plexus block is recorded at 100 Hz. The photoplethysmographic amplitude is calculated by subtracting the valley amplitude from the peak amplitude of one heartbeat in photoplethysmographic waveform. Using all the photoplethysmographic amplitudes between 0 and 25 minutes after the introduction of a block needle, a sigmoid Emax model is built. From the model, the time point, when 90% of maximum photoplethysmographic amplitude is achieved, can be derived.
Time to achieve 95% of maximum photoplethysmographic amplitude measured from the 1st finger | 25 minutes after the introduction of a block needle
  During the whole study period, the photoplethysmographic waveform obtained from the 1st and 5th fingers ipsilateral to interscalene brachial plexus block is recorded at 100 Hz. The photoplethysmographic amplitude is calculated by subtracting the valley amplitude from the peak amplitude of one heartbeat in photoplethysmographic waveform. Using all the photoplethysmographic amplitudes between 0 and 25 minutes after the introduction of a block needle, a sigmoid Emax model is built. From the model, the time point, when 95% of maximum photoplethysmographic amplitude is achieved, can be derived.
Time to achieve 99% of maximum photoplethysmographic amplitude measured from the 1st finger | 25 minutes after the introduction of a block needle
  During the whole study period, the photoplethysmographic waveform obtained from the 1st and 5th fingers ipsilateral to interscalene brachial plexus block is recorded at 100 Hz. The photoplethysmographic amplitude is calculated by subtracting the valley amplitude from the peak amplitude of one heartbeat in photoplethysmographic waveform. Using all the photoplethysmographic amplitudes between 0 and 25 minutes after the introduction of a block needle, a sigmoid Emax model is built. From the model, the time point, when 99% of maximum photoplethysmographic amplitude is achieved, can be derived.
Baseline blood flow measured from the brachial artery ipsilateral to interscalene brachial plexus block | 15 minutes before the introduction of a block needle
  The linear ultrasound transducer is placed parallel with the brachial artery at the antecubital fossa. Using pulse wave Doppler ultrasound, time velocity integral per heartbeat is calculated. The cross-sectional diameter of the artery is measured with the transducer placed transversely to the artery. The blood flow of the artery (ml/min) is the product of the averaged time velocity integral (cm), cross-sectional area of the artery (cm2), and heart rate (beats/min).
Baseline blood flow measured from the radial artery ipsilateral to interscalene brachial plexus block | 15 minutes before the introduction of a block needle
  The linear ultrasound transducer is placed parallel with the radial artery at the distal forearm area. Using pulse wave Doppler ultrasound, time velocity integral per heartbeat is calculated. The cross-sectional diameter of the artery is measured with the transducer placed transversely to the artery. The blood flow of the artery (ml/min) is the product of the averaged time velocity integral (cm), cross-sectional area of the artery (cm2), and heart rate (beats/min).
Baseline blood flow measured from the ulnar artery ipsilateral to interscalene brachial plexus block | 15 minutes before the introduction of a block needle
  The linear ultrasound transducer is placed parallel with the ulnar artery at the distal forearm area. Using pulse wave Doppler ultrasound, time velocity integral per heartbeat is calculated. The cross-sectional diameter of the artery is measured with the transducer placed transversely to the artery. The blood flow of the artery (ml/min) is the product of the averaged time velocity integral (cm), cross-sectional area of the artery (cm2), and heart rate (beats/min).
Post-block blood flow measured from the brachial artery ipsilateral to interscalene brachial plexus block | 25 minutes after the introduction of a block needle
  The linear ultrasound transducer is placed parallel with the brachial artery at the antecubital fossa. Using pulse wave Doppler ultrasound, time velocity integral per heartbeat is calculated. The cross-sectional diameter of the artery is measured with the transducer placed transversely to the artery. The blood flow of the artery (ml/min) is the product of the averaged time velocity integral (cm), cross-sectional area of the artery (cm2), and heart rate (beats/min).
Post-block blood flow measured from the radial artery ipsilateral to interscalene brachial plexus block | 25 minutes after the introduction of a block needle
  The linear ultrasound transducer is placed parallel with the radial artery at the distal forearm area. Using pulse wave Doppler ultrasound, time velocity integral per heartbeat is calculated. The cross-sectional diameter of the artery is measured with the transducer placed transversely to the artery. The blood flow of the artery (ml/min) is the product of the averaged time velocity integral (cm), cross-sectional area of the artery (cm2), and heart rate (beats/min).
Post-block blood flow measured from the ulnar artery ipsilateral to interscalene brachial plexus block | 25 minutes after the introduction of a block needle
  The linear ultrasound transducer is placed parallel with the ulnar artery at the distal forearm area. Using pulse wave Doppler ultrasound, time velocity integral per heartbeat is calculated. The cross-sectional diameter of the artery is measured with the transducer placed transversely to the artery. The blood flow of the artery (ml/min) is the product of the averaged time velocity integral (cm), cross-sectional area of the artery (cm2), and heart rate (beats/min).
Sensory blockade of the C5 dermatome | 30 minutes after the introduction of a block needle
  Using an alcohol swab, the sensory blockade of each dermatome is graded as 0 (no cold sensation), 1 (reduced cold sensation), 2 (normal cold sensation).
Sensory blockade of the C6 dermatome | 30 minutes after the introduction of a block needle
  Using an alcohol swab, the sensory blockade of each dermatome is graded as 0 (no cold sensation), 1 (reduced cold sensation), 2 (normal cold sensation).
Sensory blockade of the C7 dermatome | 30 minutes after the introduction of a block needle
  Using an alcohol swab, the sensory blockade of each dermatome is graded as 0 (no cold sensation), 1 (reduced cold sensation), 2 (normal cold sensation).
Sensory blockade of the C8 dermatome | 30 minutes after the introduction of a block needle
  Using an alcohol swab, the sensory blockade of each dermatome is graded as 0 (no cold sensation), 1 (reduced cold sensation), 2 (normal cold sensation).
Sensory blockade of the T1 dermatome | 30 minutes after the introduction of a block needle
  Using an alcohol swab, the sensory blockade of each dermatome is graded as 0 (no cold sensation), 1 (reduced cold sensation), 2 (normal cold sensation).
Motor blockade of shoulder abduction | 30 minutes after the introduction of a block needle
  Motor blockade is assessed by rating the force of movement corresponding to each nerve as 0 (complete block), 1 (partial block), or 2 (no block).
Motor blockade of elbow flexion | 30 minutes after the introduction of a block needle
  Motor blockade is assessed by rating the force of movement corresponding to each nerve as 0 (complete block), 1 (partial block), or 2 (no block).
Motor blockade of forearm supination | 30 minutes after the introduction of a block needle
  Motor blockade is assessed by rating the force of movement corresponding to each nerve as 0 (complete block), 1 (partial block), or 2 (no block).
Motor blockade of forearm pronation | 30 minutes after the introduction of a block needle
  Motor blockade is assessed by rating the force of movement corresponding to each nerve as 0 (complete block), 1 (partial block), or 2 (no block).
Motor blockade of finger abduction | 30 minutes after the introduction of a block needle
  Motor blockade is assessed by rating the force of movement corresponding to each nerve as 0 (complete block), 1 (partial block), or 2 (no block).
Motor blockade of thumb abduction | 30 minutes after the introduction of a block needle
  Motor blockade is assessed by rating the force of movement corresponding to each nerve as 0 (complete block), 1 (partial block), or 2 (no block).
Motor blockade of thumb adduction | 30 minutes after the introduction of a block needle
  Motor blockade is assessed by rating the force of movement corresponding to each nerve as 0 (complete block), 1 (partial block), or 2 (no block).
Motor blockade of thumb opposition | 30 minutes after the introduction of a block needle
  Motor blockade is assessed by rating the force of movement corresponding to each nerve as 0 (complete block), 1 (partial block), or 2 (no block).
Baseline pupil diameter ipsilateral to interscalene brachial plexus block | 5 minutes before the introduction of a block needle
  Three minutes after the adaptation in low mesopic conditions, the pupil diameter is measured for 2 seconds at 30 Hz using a portable pupillometer. The pupil diameter is obtained by averaging 60 measurement values.
Baseline pupil diameter contralateral to interscalene brachial plexus block | 5 minutes before the introduction of a block needle
  Three minutes after the adaptation in low mesopic conditions, the pupil diameter is measured for 2 seconds at 30 Hz using a portable pupillometer. The pupil diameter is obtained by averaging 60 measurement values.
Post-block pupil diameter ipsilateral to interscalene brachial plexus block | 35 minutes after the introduction of a block needle
  Three minutes after the adaptation in low mesopic conditions, the pupil diameter is measured for 2 seconds at 30 Hz using a portable pupillometer. The pupil diameter is obtained by averaging 60 measurement values.
Post-block pupil diameter contralateral to interscalene brachial plexus block | 35 minutes after the introduction of a block needle
  Three minutes after the adaptation in low mesopic conditions, the pupil diameter is measured for 2 seconds at 30 Hz using a portable pupillometer. The pupil diameter is obtained by averaging 60 measurement values.
Pain upon a pinch at the skin area for posterior portal placement (1.5-3 cm inferior and medial to the posterolateral tip of the acromion) | 1 minute before the surgical incision
  The pain intensity is rated as 0 (no pain), 1 (mild pain), and 2 (severe pain).
Pain upon surgical incision (1.5-3 cm inferior and medial to the posterolateral tip of the acromion) | An average of 1 hour after the introduction of a block needle
  The pain intensity is rated as 0 (no pain), 1 (mild pain), and 2 (severe pain).
Pain upon posterior portal placement (1.5-3 cm inferior and medial to the posterolateral tip of the acromion) | 1 minute after surgical incision
  The pain intensity is rated as 0 (no pain), 1 (mild pain), and 2 (severe pain).

OTHER OUTCOMES:
Complications related to interscalene brachial plexus block | 35 minutes after the introduction of a block needle
  Accidental puncture of the common carotid, subclavian, or vertebral artery, pneumo/hemothorax, epidural or intrathecal injection of local anesthetic, local anesthetic systemic toxicity, and other neurological complications
Baseline systolic blood pressure | 5 minutes before the introduction of a block needle
  Measured with a non-invasive blood pressure cuff
Post-block systolic blood pressure | 35 minutes after the introduction of a block needle
  Measured with a non-invasive blood pressure cuff
Baseline heart rate | 5 minutes before the introduction of a block needle
  Measured from electrocardiogram
Post-block heart rate | 35 minutes after the introduction of a block needle
  Measured from electrocardiogram

CONTACTS AND LOCATIONS:
Overall Officials: Jonghae Kim, M.D., Principal Investigator — Daegu Catholic University School of Medicine, Daegu, Republic of Korea
Locations (1):
- Daegu Catholic University Medical Center, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: No
The data will be provided upon reasonable requests to the principal investigator.